CLINICAL TRIAL: NCT01184586
Title: Dupuytren's Disease and Extracorporeal Shockwave Therapy (DupuyShock-2010) - a Randomized Trial
Brief Title: Dupuytren's Disease and Extracorporeal Shockwave Therapy (DupuyShock-2010)
Acronym: DupuyShock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Karsten Knobloch, Prof. Dr. Karsten Knobloch, FACS, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DupuyShock-2010
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Dupuytren Contracture
Keywords: function; DASH; MHQ; pain; strength
MeSH Terms: conditions — Dupuytren Contracture; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm - ESWT Storz Duolith high energy (Active Comparator): Three weekly sessions of extracorporeal shockwave therapy with focussed shock waves (STORZ DUOLITH, 1000 impulses, 0.55-0,8mJ/mm2)
  Interventions: Device: Intervention - ESWT Storz Duolith high energy
- Control - SHAM ESWT STORZ DUOLITH [0.01mJ/mm2] (Sham Comparator): Three weekly sessions of sham extracorporeal shock wave with modified probe without shockwave transduction (1000 impulses)
  Interventions: Device: CONTROL SHAM-ESWT Storz Duolith [0.01mJ/mm2]

INTERVENTIONS:
Device: Intervention - ESWT Storz Duolith high energy — Three weekly sessions of extracorporeal shockwave therapy with focussed shock waves (2000 impulses, 0,35-1,25mJ/mm2)
  Arms: Intervention arm - ESWT Storz Duolith high energy
Device: CONTROL SHAM-ESWT Storz Duolith [0.01mJ/mm2] — Three weekly sessions of sham extracorporeal shock wave (2000 impulses, 0,01mJ/mm2)
  Arms: Control - SHAM ESWT STORZ DUOLITH [0.01mJ/mm2]

SUMMARY:
Dupuytren's disease is a progressive disease due to unknown causal agents or genetics.

Dupuytren's disease contains nodules and cords in the fascia as the epicenter of disease progression. Nodules contain whorls of collagen bundles and are densely packed with contractile fibroblasts and myofibroblasts. These highly contractile cells are linked to the fascia matrix through transmembrane integrin receptors. The cytoplasmic tail domains of the alpha beta integrin receptors provide a structural link between extracellular matrix and the actomyosin cytoskeleton.

Complications of surgical partial or total aponeurectomy in Dupuytren's disease are reported in up to 10% of cases . Often, surgical complications lead to compromised flexion limiting grasping function of the involved hand . A recent 20-year-review of the literature included 41 clinical trials with complication rates reported from 3.6%to 39.1% . 16% major complications occurred with 3% digital nerve injuries, digital artery injuries in 2%, infections in 2%, and complex regional pain syndrome in 6%. Besides selective or total aponeurectomy, soft-tissue distraction has been suggested using either pneumatic devices or external fixateur .

Non-invasive options include percutaneous fasciotomy or collagenase injection. The latter has been tested in a randomized-controlled trial published in the New England Journal of Medicine with 308 patients enrolled (NCT00528606) . Collagenase clostridium histolyticum significantly reduced contractures and improved the range of motion in joints affected by advanced Dupuytren's disease. In the long-term the cords at the level of the proximal interphalangeal joint appear to more recurrent than at the metacarpophalangeal joint after collagenase injection with an eight year follow-up .

In early stage Dupuytren's contracture, radiotherapy has been suggested to limit disease progression. A cohort study of 135 patients with 208 hands involved received orthovoltage radiotherapy with a total dose of 30Gray separated by a six to eight week interval . After a follow-up of 13 years nodules and cords remained stable in 59%, improved in 10% and progressed in 31%.

Beside Dupuytren's disease, there are a number of further less common fibromatosis, such as knuckle pads, M. Ledderhose , of the plantar fascia and peyronie disease at the penis. The latter has been treated by extracorporeal shockwave therapy. A randomized-controlled trial using 2000 focused shock waves reduced pain significantly and improved erectile function and quality of life . About half of the patients in one series of 44 patients had a significant reduction in angulation following shockwave therapy .

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are patients aged 18 or over and 80 or younger
* Dupuytren's disease of stage 1-4 involving one or more fingers or the palm only

Exclusion Criteria:

* Exclusion criteria are suspected or evident pregnancy
* no Dupuytren's disease
* evident ulcerations
* no informed consent
* age under 18 years or above 80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Score of Michigan Hand Outcome Questionnaire (MHQ) [0=poor, 100= perfect] | 12 weeks
  The MHQ is a side-specific questionnaire with 25 unilateral and 12 bilateral questions, including hand function, work performance, and cosmetic appearance. It generates a score from 0 (poor) to 100 (no disability at all). The MHQ is responsive to clinical change. We have performed a validated standardized language adoption of the English MHQ into German, published in Plastic Reconstructive Surgery (Knobloch K et al. PRS 2010 in press).

SECONDARY OUTCOMES:
DASH Score [0=perfect, no impairment, 100=worst] | 12 weeks
  The DASH is a 30-item patient-reported questionnaire with two adjuncts, DASH-Sport (4 items) and DASH-Work (4-items). Notably, the validation of the aformentioned DASH score included patients suffering from Dupuytren's disease. Longitudinal construct validity has been assessed in patients including those with Dupuytren's disease and the responsiveness is moderate (effect size 0,5). The DASH questionnaire has a good validity with the subscale of SF-36 . The test-retest reliability of the DASH questionnaire has been found to be excellent (ICC = 0.96) .
Range of motion [ROM°] | 12 weeks
  Range of motion (ROM) measured in [°] using a goniometer
Grip strength [JAMAR] | 12 weeks
  Hand grip strength [kg] using a JAMAR dynanometer in three repetitions on each hand with elbow totally extended (0° flexion) and 90° flexion

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Knobloch, MD, Principal Investigator — Hannover Medical School, Germany; Peter M Vogt, MD, PhD, Study Chair — Hannover Medical School, Germany
Locations (1):
- Hannover Medical School, Plastic, Hand and Reconstructive Surgery, Hanover, Germany

REFERENCES:
- [Background] Knobloch K, Kuehn M, Papst S, Kraemer R, Vogt PM. German standardized translation of the michigan hand outcomes questionnaire for patient-related outcome measurement in Dupuytren disease. Plast Reconstr Surg. 2011 Jul;128(1):39e-40e. doi: 10.1097/PRS.0b013e318218fd70. No abstract available. PMID 21701313
- [Background] Knobloch K, Redeker J, Vogt PM. Antifibrotic medication using a combination of N-acetyl-L-cystein (NAC) and ACE inhibitors can prevent the recurrence of Dupuytren's disease. Med Hypotheses. 2009 Nov;73(5):659-61. doi: 10.1016/j.mehy.2009.08.011. Epub 2009 Sep 1. PMID 19726137
- [Background] Knobloch K, Kuehn M, Vogt PM. Focused extracorporeal shockwave therapy in Dupuytren's disease--a hypothesis. Med Hypotheses. 2011 May;76(5):635-7. doi: 10.1016/j.mehy.2011.01.018. Epub 2011 Feb 1. PMID 21277691
- [Derived] Knobloch K, Hellweg M, Sorg H, Nedelka T. Focused electromagnetic high-energetic extracorporeal shockwave (ESWT) reduces pain levels in the nodular state of Dupuytren's disease-a randomized controlled trial (DupuyShock). Lasers Med Sci. 2022 Feb;37(1):323-333. doi: 10.1007/s10103-021-03254-9. Epub 2021 Jan 23. PMID 33483776